CLINICAL TRIAL: NCT04656041
Title: A Phase II Study of Neoadjuvant NAPOX Followed by Chemoradiation With Paclitaxel and Carboplatin in Locally Advanced Esophagogastric Cancer
Brief Title: Folfox+Irinotecan+Chemort In Esophageal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Principal Investigator, Jennifer Wo, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-452
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Gastroesophageal Junction Adenocarcinoma; Esophagogastric Cancer
Keywords: Gastroesophageal Junction Adenocarcinoma; Esophagogastric cancer
MeSH Terms: interventions — Folfox protocol; irinotecan sucrosofate; Paclitaxel; Albumin-Bound Paclitaxel; Carboplatin; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- FOLFOX/ nal-IRI (Experimental): Treatment will be administered on an outpatient basis.
  * FOLFOX with nal-IRI for eight two-week cycles (16 weeks total)
  * Chemoradiation with proton or photon radiation therapy concurrent with weekly Paclitaxel and Carboplatin for 5 weeks
  * Surgery
  Interventions: Drug: FOLFOX/ nal-IRI; Drug: Paclitaxel; Drug: Carboplatin; Radiation: Proton Radiation Therapy

INTERVENTIONS:
Drug: FOLFOX/ nal-IRI — A cycle will be two weeks (14 days) long, with FOLFOX/ nal-IRI administered on days 1-3.
  The order of FOLFOX/ nal-IRI administration is as follows:
  * 1) Liposomal Irinotecan free base via IV, predetermined dosage per protocol
  * 2) Oxaliplatin via IV, predetermined dosage per protocol
  * 3) Leucovorin via IV, predetermined dosage per protocol
  * 4) 5-Fluorouracil via IV, predetermined dosage per protocol
Drug: Paclitaxel — Paclitaxel and Carboplatin will be given concurrently with radiation therapy weekly (+/- 1 day).
  Other Names: Abraxane®.
Drug: Carboplatin — Paclitaxel and Carboplatin will be given concurrently with radiation therapy weekly (+/- 1 day).
  Other Names: Paraplatin
Radiation: Proton Radiation Therapy — Chemoradiation with proton or photon radiation therapy concurrent with weekly Paclitaxel and Carboplatin for 5 weeks

SUMMARY:
In this research study, is studying how Liposomal Irinotecan in combination with the standard of care interventions FOLFOX, carboplatin paclitaxel, and radiation therapy affect gastroesophageal junction or esophagogastric cancer

This research study involves the following study intervention:

- Liposomal irinotecan

DETAILED DESCRIPTION:
The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

This research study involves the following standard of care interventions:

* FOLFOX (leucovorin calcium, 5-Fluorouracil, and oxaliplatin)
* Carboplatin
* Paclitaxel
* Radiation therapy

This research study involves the following study intervention:

- Liposomal irinotecan

It is expected that about 40 people will take part in this research study.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied. The U.S. Food and Drug Administration (FDA) has not approved liposomal irinotecan for your specific disease but it has been approved for other uses. The FDA has approved FOLFOX, carboplatin, and paclitaxel as treatment options for this disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all the following criteria in order to be eligible to participate in the study:
* Histologically or cytologically confirmed T 3/4 or N+ (> 1 cm in size or FDG avid) Siewart 1-3 gastroesophageal (GE) junction or esophagogastric cancer. Diagnosis must be confirmed by a DF/HCC institution pathology department prior to registration.
* Age 18 years or older. There will be no upper age restriction.
* ECOG performance status ≤ 1
* Life expectancy of greater than 3 months
* Participants must have adequate organ and marrow function as defined below:

  * absolute neutrophil count ≥ 1,500 cells/mm3
  * platelets ≥ 75,000 cells/mm3
  * total bilirubin ≤ 1.5 x upper limit of normal OR for patients who have undergone biliary stenting, total bilirubin of ≤ 2.0 x upper limit of normal OR two down trending values.
  * AST(SGOT) ≤ 2.5 x upper limit of normal
  * ALT (SGPT) ≤ 2.5 x upper limit of normal
  * creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 30 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* The effects of both radiation therapy and the chemotherapy agents used in this trial are known to be teratogenic. Therefore, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation plus 30 days from the last date of study drug administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Female subject of childbearing potential should have a negative urine or serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who fulfill any of the following criteria will be excluded from the study:
* Evidence of metastatic disease as determined by chest CT scan, abdomen/pelvis CT scan (or MRI with gadolinium and/or manganese) within six weeks of study entry. Distant nodal disease is allowed if it is in the radiation port.
* Any prior chemotherapy, targeted/biologic therapy, or radiation for treatment of the participant's esophagogastric cancer.
* Treatment of other invasive carcinomas within the last five years with greater than 5% risk of recurrence at time of eligibility screening. Carcinoma in-situ and basal cell carcinoma/ squamous cell carcinoma of the skin are allowed.
* Receipt of any other investigational agents within 4 weeks preceding the start of study treatment.
* Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator), such as significant cardiac or pulmonary morbidity (e.g.congestive heart failure, symptomatic coronary artery disease and/or cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months, or ongoing infection as manifested by fever.
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance or drug intake.
* Pregnant women are excluded from this study because radiation therapy and the chemotherapy agents to be used have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued while the mother is receiving protocol therapy.
* Major surgery, excluding laparoscopy, within 4 weeks of the start of study treatment, without complete recovery.
* No concurrent administration of cimetidine (as it can decrease the clearance of 5-FU). Another H2-blocker or proton pump inhibitor may be substituted before study entry.
* Known, existing uncontrolled coagulopathy.
* Prior systemic fluoropyrimidine therapy (unless given in an adjuvant setting and at least six months earlier). Prior topical fluoropyrimidine use is allowed.
* Known hypersensitivity to 5-fluorouracil or known DPD deficiency.
* History of allergic reaction(s) attributed to compounds of similar chemical or biologic composition to 5-fluorouracil, irinotecan, or oxaliplatin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response Rate | 38 Weeks
  All patients will undergo a full pathological review of their surgical specimen according to the AJCC Staging Classification, 6th. Initial gross evaluation and identification of resection margins will be performed jointly by the surgeon and the pathologist. Pathological complete response will be defined as the absence of any viable tumor cells within the pathologic specimen.

SECONDARY OUTCOMES:
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v5.0 | first dose of protocol therapy until 5 years after the end of protocol therapy
  Toxicity associated with neoadjuvant FOLFOX/ nal-IRI and chemoradiation will be summarized by category and grade according to the CTCAE version 5.0 Acute and late toxicities will be scored using Common Toxicity Criteria (CTCAE) version 5.
  Toxicities will be noted and recorded in protocol-specific case reports from the time of first dose of protocol therapy until 5 years after the end of protocol therapy
Clinical Response | 8 Weeks
  The rate of objective clinical response to induction FOLFOX/ nal-IRI and chemoradiation will be reported as the proportion of eligible patients starting protocol therapy who achieve a complete or partial response as the best overall response
Clinical Response | 16 Weeks
  The rate of objective clinical response to induction FOLFOX/ nal-IRI and chemoradiation will be reported as the proportion of eligible patients starting protocol therapy who achieve a complete or partial response as the best overall response
Clinical Response | 25 Weeks
  The rate of objective clinical response to induction FOLFOX/ nal-IRI and chemoradiation will be reported as the proportion of eligible patients starting protocol therapy who achieve a complete or partial response as the best overall response
Progression-Free Survival (PFS) | duration from the first date of protocol therapy to the earliest date of disease progression up 5 years
  Progression-free survival (PFS) is defined as the duration from the first date of protocol therapy to the earliest date of disease progression per RECIST criteria or death due to any cause. PFS time will be censored at the date of last follow-up for patients still alive with no documentation of progressive disease. The PFS rate will be estimated using the Kaplan-Meier method with 95% confidence intervals based on the complementary log-log transformation.
Overall Survival | first date of protocol therapy to the date of death due to any cause and will be censored at the date of last follow-up for patients still alive up to 5 years
  Overall survival (OS) is defined as the duration from the first date of protocol therapy to the date of death due to any cause and will be censored at the date of last follow-up for patients still alive. The OS rate will be estimated using the Kaplan-Meier method with 95% confidence intervals based on the complementary log-log transformation

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wo, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth-Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital at Newton Wellesley Hospital, Newton, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation